CLINICAL TRIAL: NCT06858748
Title: Canadian Consortium for Understanding the Role of Airway Mucus Occlusions in Asthma, COPD and Chronic Cough
Brief Title: Canadian Consortium on Airway Mucus Occlusions in Asthma, COPD and Chronic Cough
Acronym: CANMuc
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: CANMuc01
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD); Chronic Cough (CC)
Keywords: mucus occlusions; asthma; Chronic Cough (CC); Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Chronic Cough | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, PBMC, sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Asthma
  Interventions: Other: Observational
- Chronic Obstructive Pulmonary Disease (COPD)
  Interventions: Other: Observational
- Chronic cough
  Interventions: Other: Observational
- Control group
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This is a 24-month observational study in adults in three disease domains, consisting of screening visit, baseline visit, quarterly telemonitoring visit and end of monitoring period

SUMMARY:
Chronic lung diseases affect one in five Canadians, causing symptoms such as cough, breathlessness, and wheeze. Despite advancements in medical care, these conditions not only impact individuals and their close circles but also present substantial clinical and economic challenges at a national level. This grant is dedicated to addressing three prevalent lung diseases: asthma, chronic obstructive pulmonary disease (COPD), and chronic cough. An alliance of clinicians, scientists, knowledge users, and patient partners from across Canada have come together to establish the Canadian Consortium for Understanding the Role of Airway Mucus Occlusions in Asthma, COPD, and Chronic Cough - "CANMuc." Mucus plays a pivotal role in the symptoms and severity of lung diseases, but its clinical assessment has been challenging. Fortunately, recent medical advances, particularly chest computed tomography (CT), facilitate visualizing and quantifying mucus in patients with lung diseases. Our goal is to initially assess mucus plugging in a diverse group of Canadians without lung disease and then compare these findings to those with asthma, COPD, and chronic cough. The investigators will recruit 100 healthy volunteers for comprehensive clinical and research evaluations, including sputum analyses, breathing tests, quality of life assessments, cough monitoring, and CT scans. In addition, testing will be conducted twice, two years apart, in 240 adult and 50 pediatric participants. This approach will enable the investigators to understand the burden of mucus and how it changes over time, explore proteins or chemicals in mucus that predict mucus persistence, and identify biomarkers that can help guide physicians to prescribe targeted treatments that might work better than others. The CANMuc team's findings will guide strategies for identifying and treating mucus plugging, inform policymakers, and share knowledge with Canadians living with asthma, COPD, and chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (≥18 years old)

Asthma: Respiratory physician confirmed diagnosis of moderate-to-severe asthma and Historical objective evidence of asthma and/or specialist/respirologist confirmation (post-bronchodilator reversibility and/or methacholine bronchoprovocation test <8 mg/mL)

COPD: Respiratory physician confirmed diagnosis of COPD that is moderate-to-severe according to GOLD criteria (post-bronchodilator FEV1/FVC<LLN and FEV1< 80%pred) and CAT score ≥10 or mMRC score ≥ 2

Chronic cough: Refractory Chronic Cough (RCC) and Unexplained Chronic Cough (UCC) lasting >1 year with Normal chest radiograph and no airflow obstruction (FEV1/FVC >Lower Limit of Normal)

Healthy participants: No history of respiratory disease or other pulmonary disorders and no use of inhaled medications or corticosteroids with normal spirometry and Modified Medical Research Council (mMRC) Dyspnea Scale =<1

Exclusion Criteria:

* Pregnant or breastfeeding
* Current smoker or >10 yr pack history or smoked within the last 6 months
* Exacerbation within 4 weeks of recruitment
* Preterm birth (≤36 weeks gestation) or perinatal complications
* History of other pulmonary disorders
* Specialist/Respirologist suspects primary ciliary dyskinesia (PCD)
* Current use of mucolytic medications
* Memory, cognitive, or psychiatric limitations that may prevent optimal participation
* Treatment with current biologic therapy: anti-IgE mAb within 130 days, anti-IL-4/4R, IL-5/5R, IL-13, or TSLP within 2 months or 5 half-lives whichever is longer prior to visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A coalition of 25 clinicians and scientists from across Canada have united to establish the Canadian Consortium for understanding the role of airway mucus occlusions in chronic cough, COPD, and asthma (CANMuc).
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Computed Tomography mucus score | Baseline/Day 0 and End of Assessment/48 months
  Quantify CT mucus score and evaluate its cross-sectional and longitudinal relationship with sputum rheology and inflammatory phenotype in a healthy cohort compared to disease groups at baseline and follow-up

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Robarts Research Institute, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Quebec Heart and Lung Institute - Laval University, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided